CLINICAL TRIAL: NCT04797065
Title: Impact of 9-minute Withdrawal Time on Adenoma Miss Rate: A Multicenter, Prospective, Randomized Controlled Trial of Tandem Colonoscopy
Brief Title: 9 Minutes for Tandem Colonoscopy Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other); Yantaishan Hospital of Yantai City, Yantai, China (Unknown); Seventh Medical Center of PLA Army General Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The First Affiliated Hospital of the Medical College, Shihezi University (Unknown); Shanghai 8th People's Hospital (Other); Shanxi Provincial People's Hospital (Other Government); Qinghai People's Hospital (Other); Leqing People's Hospital (Unknown); Afﬁliated Hospital of North Sichuan Medical College (Other); Zhejiang University (Other); Songjiang Hospital Affiliated to Shanghai Jiaotong University School of Medicine (Other Government); The General Hospital of Eastern Theater Command (Other); Heilongjiang provincial hospital (Unknown); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: withdrawal time-2
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Colon Polyp; Colorectal Adenoma
Keywords: withdrawal time; adenoma miss rate; tandem colonoscopy; adenoma detection rate
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-minute then 9-minute withdrawal (Experimental): Patients in 6-minute then 9-minute withdrawal group will first be carefully observed in 6 minutes then in 9 minutes during the segmental withdrawal.
  At 6-minute withdrawal, the left colon, transverse colon and right colon will take 2 minutes each. Then at 9-minute withdrawal, the observation of the left colon, transverse colon and the right colon will be maintained for 3 minutes each.
  A stop watch will be utilized to remind endoscopists the withdrawal time. The time to perform polyp biopsy will not be included.
  Interventions: Procedure: 6-minute then 9-minute withdrawal
- 9-minute then 6-minute withdrawal (Active Comparator): Patients in 9-minute then 6-minute withdrawal group will first be carefully observed in 9 minutes then in 6 minutes during the segmental withdrawal.
  At 9-minute withdrawal, the left colon, transverse colon and right colon will take 3 minutes each. Then at 6-minute withdrawal, the observation of the left colon, transverse colon and the right colon will be maintained for 2 minutes each.
  A stop watch will be utilized to remind endoscopists the withdrawal time. The time to perform polyp biopsy will not be included.
  Interventions: Procedure: 9-minute then 6-minute withdrawal

INTERVENTIONS:
Procedure: 6-minute then 9-minute withdrawal — Patients in 6-minute then 9-minute withdrawal group will first be carefully observed in 2 minutes then in 3 minutes during each colonic segment.
  In actual performance, withdrawal of the right colon, transverse colon and the left colon can be operated in segmental tandem colonoscopy. Taking the right colon as an example, after the endoscope reaches the cecum, it can be withdrawn to the splenic curvature in 2 minutes, then reentered the cecum and withdrawn to the splenic curvature in 3 minutes.
  Arms: 6-minute then 9-minute withdrawal
Procedure: 9-minute then 6-minute withdrawal — Patients in 9-minute then 6-minute withdrawal group will first be carefully observed in 3 minutes then in 2 minutes during each colonic segment.
  In actual performance, withdrawal of the right colon, transverse colon and the left colon can be operated in segmental tandem colonoscopy. Taking the right colon as an example, after the endoscope reaches the cecum, it can be withdrawn to the splenic curvature in 3 minutes, then reentered the cecum and withdrawn to the splenic curvature in 2 minutes.
  Arms: 9-minute then 6-minute withdrawal

SUMMARY:
A mean withdrawal time of at least 6 minutes has been considered to be one of the critical quality criterions of colonoscopy. Recently, our group completed a multicenter randomized controlled trial, which proved that prolonging the withdrawal time to 9 minutes could significantly improve the adenoma detection rate of colonoscopists, especially for young colonoscopists and proximal colon. However, it has some limitations in included participates (mixed indications for colonoscopy) and cannot illustrate the impact of withdrawal time on adenoma miss rate in a parallel randomized design. It is necessary to include tandem colonoscopy and adopt strict criteria of the screening population to confirm the effect of the 9-minute withdrawal time on the adenoma miss rate. Therefore, the investigators plan to conduct a multicenter, randomized controlled trial of tandem colonoscopy to compare adenoma miss rate of 6-minute and 9-minute withdrawal in screening population.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is between 40-75.
* Patients who have indications for screening
* Patients who have signed inform consent form.

Exclusion Criteria:

* Patients who have undergone colonic resection or polypectomy
* Patients with alarming signs and symptoms of colorectal cancer: hematochezia, melena, anemia, weight loss, abdominal mass, positive digital rectal examination
* Patients with abnormal blood coagulation or taking antiplatelets or anticoagulants within 7 days
* Patients with inflammatory bowel diseases
* Patients with a history of abdominal surgery, or highly suspected or confirmed colorectal cancers by radiographic and laboratory tests
* Patients with hereditary colorectal cancer syndrome (including familial adenomatous polyposis).
* Patients with pregnancy, severe chronic cardiopulmonary and renal disease.
* Patients with failed cecal intubation
* Patients with poor BPQ that necessitated a second bowel preparation
* Patients with therapeutic colonoscopy for existing lesions
* Patients refusing to participate or to provide informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
adenoma miss rate(AMR) | 60 minutes
  Adenomas detected in the second-pass examination were defined as missed adenomas; the AMR was defined as follows: number of adenomas detected in the second-pass examination/total number of adenomas detected in the two pass.

SECONDARY OUTCOMES:
advanced adenoma miss rate(AAMR) | 60 minutes
  AAMR is the number of advanced adenomas detected in the second-pass examination/total number of advanced adenomas detected in the two pass.
adenoma detection rate(ADR) | 60 minutes
  ADR is the number of patients with at least one adenoma, divided by the total number of patients.
adenomas per colonoscopy(APC) | 60 minutes
  APC was calculated as the number of adenomas detected during colonoscopy withdraw divided by the number of colonoscopies.
patient-level AMR(pAMR) | 60 minutes
  the number of participants with adenomas detected only during the second-pass colonoscopy divided by the total number of participants with adenomas detected during the tandem colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Background] Zhao S, Yang X, Wang S, Meng Q, Wang R, Bo L, Chang X, Pan P, Xia T, Yang F, Yao J, Zheng J, Sheng J, Zhao X, Tang S, Wang Y, Wang Y, Gong A, Chen W, Shen J, Zhu X, Wang S, Yan C, Yang Y, Zhu Y, Ma RJ, Wang R, Ma Y, Li Z, Bai Y. Impact of 9-Minute Withdrawal Time on the Adenoma Detection Rate: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e168-e181. doi: 10.1016/j.cgh.2020.11.019. Epub 2020 Nov 19. PMID 33220526
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Derived] Zhao S, Song Y, Wang S, Wang R, Feng Z, Gong A, Yang X, Pan P, Yao D, Zhang J, Zhu Y, Li T, Bi J, Ren X, Tang X, Li Q, Yu D, Zheng J, Song B, Wang P, Chen W, Shang G, Xu Y, Xu P, Lai Y, Xu H, Yang X, Sheng J, Tao Y, Li X, Zhu Y, Zhang X, Shen H, Ma Y, Wang F, Wu L, Wang X, Li Z, Bai Y. Reduced Adenoma Miss Rate With 9-Minute vs 6-Minute Withdrawal Times for Screening Colonoscopy: A Multicenter Randomized Tandem Trial. Am J Gastroenterol. 2023 May 1;118(5):802-811. doi: 10.14309/ajg.0000000000002055. Epub 2022 Oct 11. PMID 36219172